CLINICAL TRIAL: NCT04598503
Title: Prevalence, Types and Risk Factors of Congenital Anomalies(A Hospital Based Study)
Brief Title: Congenital Anomalies and Risk Factors
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Shalaby, principal investigator, Assiut University
Other Study IDs: Assiut University CH
Record Dates: First submitted 2020-10-11; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Congenital Anomalies
MeSH Terms: conditions — Congenital Abnormalities | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: All the babies admitted to the hospital with congenital anomalies during this period were included
  Interventions: Other: full history and clinical examination
- control: newborns without congenital anomalies
  Interventions: Other: full history and clinical examination

INTERVENTIONS:
Other: full history and clinical examination — For each case, a detailed perinatal and maternal and family history were obtained by interviewing questionnaire. Diagnosis of congenital anomalies was based on clinical evaluation of newborn babies by the neonatologist and other appropriate investigations such as radiography, ultrasonography, echocardiography and chromosomal analysis etc... Classification of anomalies is done by systems according to WHO international classification of diseases (ICD10) [10]. Data was entered into excel data sheet and appropriate statistical analysis was performed. The prevalence was calculated by dividing the number of CA during the 6 months (173) by the total number of admission during this period (753).

SUMMARY:
The aim of the study is to determine the prevalence, describe the types and risk factors of congenital anomalies among newborns admitted to Neonatal Intensive Care Unit (NICU) of Assiut University Children Hospital (AUCH). It is a prospective and a case control study was performed and screening of the newborn admitted at NICU of Assiut University Children Hospital during the period of 6 months from 1-12-2017 to the end of 5-2018 the sample was 346 newborns, 173 cases and 173 control. Data were collected using a record checklist and an interviewing questionnaire. Conclusion: The prevalence of congenital anomalies was 22.97%. The most common anomalies were gastrointestinal anomalies (GIT), musculoskeletal anomalies, multiple anomalies and circulatory system anomalies. The risk factors were consanguineous marriage, positive family history, urban areas, full-term and singleton pregnancies.

DETAILED DESCRIPTION:
The aim of the study is to determine the prevalence, describe the types and risk factors of congenital anomalies among newborns admitted to Neonatal Intensive Care Unit (NICU). Study design: This is a prospective case control study was carried out in the neonatal intensive care unit. It is a tertiary care center. The center provides multi-specialist care and serves as a major referral center for hospitals within and outside the city. The study was done during the period of 6 months from December 2017 to May 2018. Patients: All the babies admitted to the hospital with congenital anomalies during this period were included. All stillbirths were excluded from this study. The sample was 346 newborns, 173 cases and 173 control. For each case, a detailed perinatal and maternal and family history were obtained by interviewing questionnaire. Diagnosis of congenital anomalies was based on clinical evaluation of newborn babies by the neonatologist and other appropriate investigations such as radiography, ultrasonography, echocardiography and chromosomal analysis etc... Classification of anomalies is done by systems according to WHO international classification of diseases (ICD10) [10]. Data was entered into excel data sheet and appropriate statistical analysis was performed. The prevalence was calculated by dividing the number of CA during the 6 months (173) by the total number of admission during this period (753). Statistical analysis: Data were analyzed using (SPSS Statistics for Windows, Version 21.0, NY). Descriptive analysis of the whole sample; where data were expressed as mean values and standard deviations for quantitative variables, and numbers and frequencies for qualitative variables. Bivariate analysis was performed to assess associations between various independent variables and the dependent variable (presence of congenital anomalies), chi-square was used to compare the difference in distribution of frequencies among different groups and if number inside the cell was small we used Fisher's Exact Test. Independent sample T-test was used to compare the difference in means among different groups. A significant p value was considered when it less than or equal 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All the babies admitted to the hospital with congenital anomalies during this period were included.

Exclusion Criteria:

* All stillbirths were excluded from this study.

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All the babies admitted to the hospital with congenital anomalies during this period were included.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
prevalence of congenital anomalies | 6months
  The prevalence was calculated by dividing the number of CA during the 6 months (173) by the total number of admission during this period (753) newborns admitted to Neonatal Intensive Care Unit (NICU)

SECONDARY OUTCOMES:
risk factors | 6months
  To determined the risk factors of congenital anomalies by a detailed perinatal, maternal and family history were obtained by interviewing questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Amira M. Shalaby, Lecturer, Principal Investigator — Assiut University Children Hospital
Locations (1):
- Assiut University Children Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Prevalence, types and risk factors of congenital anomalies